CLINICAL TRIAL: NCT03954379
Title: Opioid Sparing Analgesic Strategies for Enhanced Recovery After Total Knee Arthroplasty
Brief Title: IPACK Study in Total Knee Arthroplasty Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-5920
Record Dates: First submitted 2019-04-16; First posted 2019-05-17 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-03

CONDITIONS: Knee Replacement Arthroplasty
MeSH Terms: interventions — Standard of Care; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Block room and anesthesia staff performing nerve blocks and administering sedation will be informed to which study group patient is allocated. The patient and independent investigator carrying out follow up assessments will remain blinded to the end of the study. If the patient wishes to know the study group assignment, the patient will be informed at the end of their final 6 week follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C ( Comparator Group ) (Active Comparator): Standard of care: Adductor Canal Block(ACB), Spinal Anesthesia (SA) and Peri-op Pain management
  Interventions: Drug: Standard of Care (ACB, SA, peri-op pain management); Procedure: Periarticular Local Anesthetic Infiltration; Drug: IV Dexamethasone 8mg at the end of surgery as standard of care
- Group S ( Study Group ) (Experimental): iPACK and multi-modal analgesic regimen
  Interventions: Drug: IPACK and multi-modal analgesic regimen; Procedure: Periarticular Local Anesthetic Infiltration; Drug: IV Dexamethasone 8mg at the end of surgery as standard of care

INTERVENTIONS:
Drug: Standard of Care (ACB, SA, peri-op pain management) — INTERVENTION BEFORE SURGERY
  Adductor Canal Block will be done using Adductor canal catheter (tube in the thigh) + injection of freezing medication
  INTERVENTION DURING SURGERY
  IV propofol for sedation
  INTERVENTION AFTER SURGERY
  Injection of salty water through the tube in the thigh x 2
  Other Names: ACB
  Arms: Group C ( Comparator Group )
Drug: IPACK and multi-modal analgesic regimen — INTERVENTION BEFORE SURGERY
  1. Adductor Canal Block will be done using Adductor canal catheter (tube in the thigh) + injection of freezing medication
  2. iPACK block ( infiltration between Popliteal Artery and posterior Capsule of the Knee) - injection of freezing medication in the back of the knee
  INTERVENTION DURING SURGERY
  1. IV dexmedetomidine
  2. IV ketamine Both for sedation
  INTERVENTION AFTER SURGERY
  1. injection of freezing medication through the tube in the thigh x 2
  2. IV dexamethasone 8 mg 1 day after surgery
  Other Names: Infilteration between popliteal artery and posterior capsule of the knee
  Arms: Group S ( Study Group )
Procedure: Periarticular Local Anesthetic Infiltration — INTERVENTION DURING SURGERY
  Other Names: LAI
Drug: IV Dexamethasone 8mg at the end of surgery as standard of care — INTERVENTION DURING SURGERY
  Other Names: IV Dexamethasone Infusion

SUMMARY:
This study proposes to compare current multimodal analgesic treatment for TKA with a new multimodal analgesic regimen to demonstrate decreased opioid requirement, time to rehabilitation, and time to reach hospital discharge.

DETAILED DESCRIPTION:
Total knee replacement surgery (TKA) causes severe pain and this procedure is the most common reason patients are prescribed strong opioid drugs in hospital. As a result they are slow to begin rehabilitation after surgery, and are late in hospital discharge. Ontario hospitals are constantly challenged to meet growing demands of TKA and in fact increased demand has overcome the health care system resulting in TKA wait time (Ontario actual: 286 days vs. target: 182 days).1 One strategy to accommodate expanding volume and reduce wait time is to reduce hospital length of stay (LOS) through an enhanced recovery program.2 One essential component is further improvement of postoperative pain treatment to expedite rehabilitation and hospital discharge.

Treatment of severe post TKA pain often requires potent opioids but their excessive and prolonged use has negative consequences e.g., increased perioperative adverse events and longer LOS.3 Approximately 8% of opioid naive TKA patients become chronic opioid users at 6 months and the duration of prescription is the strongest predictor of misuse.4 Knowing that the opioid crisis in Canada is steadily growing and prescription opioids play a significant role in dependence and misuse,5 an effective perioperative opioid minimization analgesic program is mandatory for TKA patients.

Current multimodal analgesic treatment for TKA consists of oral non opioid drugs e.g., acetaminophen and non steroidal anti-inflammatory agents (NSAIDs) and surgeon performed peri-articular local anesthesia infiltration, however this is only partially effective.6 The regional analgesic effect is often short lived (< 8 hours). Failure to sustain effective analgesia necessitates continued heavy reliance on opioids.

Several new treatments have been recently described for post TKA pain. They are: IV dexamethasone (steroid),7 dexmedetomidine (alpha 2 agonist)8, ketamine (NMDA antagonist)9 and 2 novel nerve block procedures- adductor canal block10 and iPACK block (infiltration between popliteal artery and posterior capsule of the knee).11 While each individual intervention has demonstrable analgesic benefit, the impact of incorporating all new treatments into the current analgesic regimen remains unknown.

The investigators believe that the new multimodal analgesic regimen proposed in this study will significantly decrease opioid requirement, time to rehabilitation, and time to reach hospital discharge criteria. It may also decrease the duration of opioid prescription for pain relief after hospital discharge. Although investigator's preliminary experience with this new regimen in 10 patients is promising, robust evidence showing its sustained opioid sparing analgesic effect is lacking.

ELIGIBILITY:
Inclusion criteria:

* English-speaking;
* Age 18 - 85;
* BMI ≤ 38;
* Undergoing unilateral primary total knee arthroplasty surgery.

Exclusion criteria:

* inability to give informed consent
* patient refusal
* pregnancy, patients who are breastfeeding
* contraindication to nerve blocks or multimodal analgesia
* contraindication or hypersensitivity to any of the study drugs (celecoxib, acetaminophen, morphine, ropivacaine, bupivacaine, ketamine, dexmedetomidine, dexamethasone, ketorolac, epinephrine, sulfonamides)
* chronic pain disorders (> 50 mg oral morphine equivalence per day at time of recruitment)
* medical or recreational use of marijuana and substance abuse (e.g., alcoholism),
* complications after surgery that result in discharge to a location other than home
* severe cardiovascular diseases e.g., heart failure, significant dysrhythmias; uncontrolled low blood pressure e.g., systolic blood pressure ≤ 100 mm Hg while on antihypertensive medication(s)
* respiratory diseases e.g., severe asthma, urticaria, or allergic-type reactions after taking acetylsalicylic acid (ASA) or other NSAIDs; severe acute or chronic respiratory disease and obstructive airway
* severe or active liver disease
* severe inflammatory bowel disease
* severe renal impairment (creatinine clearance <30 mL/min)
* uncontrolled diabetes (type 1 or 2)
* active bleeding condition (e.g., postoperative or gastro-intestinal bleeding)
* severe psychiatric disorders and intake of monoamine oxidase inhibitors
* neurologic disorders (e.g., operative extremity neuropathy, delirium tremens, uncontrolled convulsive disorders, increased cerebrospinal or intracranial pressure)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption in MG | 24 hours
  Cumulative 24 hour oral hydromorphone and oxycodone equivalent consumption

SECONDARY OUTCOMES:
Pain scores at rest using numerical rating scale (NRS, 0 to 10) | 0-48 hours after surgery
  0, 12, 18, 24, 36 and 48 hours after surgery and also pain scores during physical therapy daily
Opioid consumption in MG | 12 hours to 6 weeks after surgery
  Analgesic consumption at 12, 18, 36 and 48 hours and 1, 2 and 6 weeks after surgery
Quality of Recovery (QoR) assessed using a validated QoR-15 tool ( Total score range- 0 to 150, higher values represent a better outcome) | Baseline, 24-hour, 48-hour and 2-weeks after surgery
  Treatment effect will be estimated using a linear regression model, with baseline QoR score as a covariate.
Time to reach physical therapy milestones in hours | 0-72 hours after surgery
  The post TKA milestones are: knee flexion ≥ 90 degrees, get in and out of bed by self, safe transfer to bathroom with or without assistance, walk with an assistive device on a level surface for a short distance and being able to climb up and down 2 or 3 stairs. steps or flights of stairs?
Time to reach hospital discharge criteria in hours | 24 to 72 hours after surgery until discharge
  The 4 criteria are: 1) adequate analgesia (numerical rating scale <4/10); 2) independence from IV opioids ≥ 12 hours; 3) ability to independently stand and sit down (evaluated with the Timed Up and Go test and 4) unassisted ambulation ≥ 30 mins (evaluated with the 6-min walk test)
Incidence of adverse events related to nerve block procedures | Post-op 24 to 72 hours
  muscle weakness, systemic toxicity
Incidence of adverse events related to opioid consumption | Post-op 24 to 72 hours
  nausea, vomiting, dizziness, sedation

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No